CLINICAL TRIAL: NCT06469671
Title: Artificial Intelligence - Assisted Colonoscopy in Diagnosis of Colorectal Neoplasms: Russian Multicenter Randomised Open - Label Trial
Brief Title: Effectiveness of Artificial Intelligence - Assisted Colonoscopy in Colorectal Neoplasms
Acronym: ArtInCol
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: State Scientific Centre of Coloproctology, Russian Federation (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 7-24
Record Dates: First submitted 2024-06-05; First posted 2024-06-21 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Colonic Neoplasms; Colonic Polyp; Diagnosis
MeSH Terms: conditions — Colonic Neoplasms; Colonic Polyps; Disease | interventions — Colonoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Artificial intelligence - assisted colonoscopy (Experimental): The decision making system based on artificial intelligence. Real - time artificial intelligence - assisted colonoscopy will be performed in this group.
  Detection of polyps is based on real time fixing a frame on the screen.
  Interventions: Device: The system based on real - time artificial intelligence - assisted for colonoscopy
- Conventional colonoscopy (Active Comparator): Conventional colonoscopy will be performed in this group
  Interventions: Device: The system based on real - time artificial intelligence - assisted for colonoscopy

INTERVENTIONS:
Device: The system based on real - time artificial intelligence - assisted for colonoscopy — Russian medical decision support system based on artificial intelligence "ArtInCol"

SUMMARY:
The primary goal of this study is to estimate the effectiveness of a medical decision support system based on artificial intelligence in the endoscopic diagnosis of benign tumors.

Researchers will compare Adenoma detection rate between "artificial intelligence - assisted colonoscopy" and "conventional colonoscopy" groups to evaluate the clinical effectiveness of artificial intelligence model.

DETAILED DESCRIPTION:
The primary outcome is adenoma detection rate per patient.

The secondary outcomes will be measured:

* Polyps detection rate (all type of lesions) per patient;
* Number of adenomas per patient;
* Number of polyps per patient;

ELIGIBILITY:
Inclusion Criteria:

* Screening coloscopy is needed

Exclusion Criteria:

* Indications for colonoscopy
* Previously detected colorectal neoplasms
* Previously performed colorectal surgery
* Colorectal cancer
* Inflammatory bowel disease

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Adenoma detection rate | during the procedure
  In each group, the percentage of patients with at least one histologically proven adenoma or carcinoma

SECONDARY OUTCOMES:
Polyps detection rate | during the procedure
  In each group, the number of patients with all type of neoplasms (polyps) was detected as a percentage of the total number of patients.
Number of polyps | during the procedure
  In each group, the number of detected all type of polyps
Number of adenomas | during the procedure
  In each group, the number of detected adenomas

CONTACTS AND LOCATIONS:
Overall Officials: Sergey Achkasov, Principal Investigator — State scientific centre of coloproctology, Moscow
Locations (1):
- Airat Mingazov, Moscow, Russia